CLINICAL TRIAL: NCT03010358
Title: A Phase I/II Study of Syk Inhibitor Entospletinib (GS-9973) in Combination With Obinutuzumab in Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) and B-Cell Malignancies
Brief Title: Entospletinib and Obinutuzumab in Treating Patients With Relapsed Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, or Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexey Danilov, MD (Other)
Collaborators: Gilead Sciences (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor-Investigator, Alexey Danilov, MD, Adjunct Associate Professor, OHSU Knight Cancer Institute
Organization: OHSU Knight Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016140; NCI-2016-02029 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00016140 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Anemia; B-Cell Prolymphocytic Leukemia; Grade 1 Follicular Lymphoma; Grade 2 Follicular Lymphoma; Grade 3a Follicular Lymphoma; Hairy Cell Leukemia; Lymphoplasmacytic Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma; Richter Syndrome
MeSH Terms: conditions — Anemia; Leukemia, Prolymphocytic, B-Cell; Lymphoma, Follicular; Leukemia, Hairy Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (entospletinib, obinutuzumab) (Experimental): Patients receive entospletinib PO either QD or BID on days -7 to -1 (run-in phase) depending on the assigned dose level. Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of the first cycle, and on day 1 of subsequent cycles. Treatment with obinutuzumab repeats every 28 days for up to 6 cycles and daily treatment with entospletinib continues every 28 days for up to 12 cycles in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Entospletinib; Other: Laboratory Biomarker Analysis; Biological: Obinutuzumab; Other: Pharmacological Study

INTERVENTIONS:
Drug: Entospletinib — Given PO
  Other Names: ENTO; GS 9973; GS-9973
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effect and best dose of entospletinib when giving together with obinutuzumab and to see how well they work in treating patients with chronic lymphocytic leukemia, small lymphocytic lymphoma, or non-Hodgkin lymphoma that has come back. Entospletinib may stop the growth of cancer cells by blocking some of the enzymes need for cell growth. Monoclonal antibodies, such as obinutuzumab, may interfere with the ability of cancer cells to grow and spread. Giving entospletinib and obinutuzumab together may work better in treating patients with chronic lymphocytic leukemia, small lymphocytic lymphoma, or non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of entospletinib administered in combination with obinutuzumab in patients with relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) and non-Hodgkin lymphoma (NHL), and identify the dose for phase 2 expansion. (Phase I) II. To evaluate the efficacy of entospletinib in combination with obinutuzumab in patients with relapsed or refractory CLL/SLL, as measured by complete response (CR) rate. (Phase II)

SECONDARY OBJECTIVES:

I. Objective response rate (ORR, defined as complete remission, complete response with incomplete marrow recovery, partial remission and nodular partial response). (Phase II) II. Event free survival defined as the interval between the date of first study treatment and the date of objective signs of disease recurrence, subsequent anti-leukemic therapy, or death, whichever is first reported. (Phase II) III. Safety and tolerability of entospletinib in combination with obinutuzumab by adverse events (AEs). (Phase II)

EXPLORATORY OBJECTIVES:

I. Peripheral blood B-cell depletion and recovery. II. Pharmacodynamics effects of in vivo administration of entospletinib on NFkappaB activation and expression of anti-apoptotic proteins in CLL cells.

III. Association of established biomarkers (chromosomal abnormalities, immunoglobulin heavy chain [IGHV] mutational status, p53 mutational status) with response (ORR and event-free survival [EFS]) to entospletinib (ENTO) in combination with obinutuzumab in patients with relapsed/refractory CLL.

OUTLINE: This is a phase I, dose-escalation study of entospletinib followed by a phase II study.

Patients receive entospletinib orally (PO) either once a day (QD) or twice a day (BID) on days -7 to -1 (run-in phase) depending on the assigned dose level. Patients also receive obinutuzumab intravenously (IV) on days 1, 2, 8, and 15 of the first cycle and on day 1 of all subsequent cycles. Treatment with obinutuzumab repeats every 28 days for up to 6 cycles and daily treatment with entospletinib continues every 28 days for up to 12 cycles in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up every 3 months for 12 months then every 6 months thereafter. In the event of study closure, patients who are receiving study drug at the time of closure will complete an abbreviated End of Treatment (EOT) visit. No additional follow up will occur.

ELIGIBILITY:
Inclusion Criteria:

* Phase I portion of the study: Histologically or flow cytometry confirmed diagnosis of B-CLL/SLL according to National Cancer Institute (NCI)-Working Group (WG) 1996 guidelines
* Phase I portion of the study: The following types of NHL as documented by medical records and with histology based on criteria established by the World Health Organization (WHO):

  * Mantle cell lymphoma (MCL)
  * Follicular lymphoma (FL) - grades 1-3a
  * Lymphoplasmacytic lymphoma (LPL)
  * Marginal zone lymphoma (MZL)
  * CLL in Richter's transformation
  * B-cell prolymphocytic leukemia
* Phase I portion of the study: Patients with histologically confirmed classical hairy cell leukemia (HCL)
* Phase II portion of the study - histologically or flow cytometry confirmed diagnosis of BCLL/SLL according to NCI-WG 1996 guidelines; patients who lack CD23 expression on their leukemia cells should be examined for (and found NOT to have) either t(11;14) or cyclin D1 overexpression, to rule out mantle cell lymphoma
* Patients underwent >= 1 prior chemotherapy-based or immunotherapy-based regimen or targeted therapy (e.g., inhibitors of BTK, PI3K etc.) administered for >= 2 cycles, and have had either documented disease progression or no response (stable disease) to the most recent treatment regimen
* Patients with CLL/SLL must demonstrate active disease meeting at least 1 of the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria for requiring treatment:

  * A minimum of any one of the following constitutional symptoms:

    * Unintentional weight loss > 10% within the previous 6 months prior to screening
    * Extreme fatigue (unable to work or perform usual activities)
    * Fevers of greater than 100.5 Fahrenheit (F) for >= 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure as manifested by the development of, or worsening of anemia or thrombocytopenia
  * Massive (i.e., > 6 cm below the left costal margin), progressive or symptomatic splenomegaly
  * Massive nodes or clusters (i.e., > 10 cm in longest diameter) or progressive lymphadenopathy
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period, or an anticipated doubling time of less than 6 months
  * Autoimmune anemia or thrombocytopenia that is poorly responsive to corticosteroids
* Patients with HCL must be intolerant of or not candidates for purine analog-based therapy, or failed to achieve response (CR or partial response [PR]) or relapsed within 2 years of such therapy, AND meet the standard treatment initiation criteria (absolute neutrophil count [ANC] =< 1000/uL, hemoglobin [Hgb] =< 10 g/dL, platelet count =< 100,000/uL); patients with indolent lymphoma (FL, LPL, MZL) and patients with B-cell prolymphocytic leukemia must have an indication for treatment in the opinion of the investigator; patients with MCL and patients with CLL in Richter's transformation should have previously received or not be candidates for high dose chemotherapy/autologous stem cell transplant
* For diseases other than CLL, LPL, and HCL, presence of radiographically measurable lymphadenopathy or extra-nodal lymphoid malignancy (defined as the presence of >= 1 lesion that measures >= 2.0 cm in the longest dimension [LD] and >= 1.0 cm in the longest perpendicular dimension [LPD] as assessed by computed tomography [CT] or magnetic resonance imaging [MRI]); for LPL, measurable disease will be defined as serum monoclonal IgM > 0.5 g/dL or meeting at least 1 of the recommendations from the Second International Workshop on LPL for requiring treatment
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Direct bilirubin =< 2 X institutional upper limit of normal (ULN) (unless due to known Gilbert's syndrome or compensated hemolysis directly attributable to CLL)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) less than 2.5 X institutional ULN
* Estimated creatinine clearance (CrCL) using the Cockcroft-Gault equation >= 50 mL/min
* Platelets >= 50,000/mm^3 independent of transfusion support, with no active bleeding
* Absolute neutrophil count (ANC) >= 1000/mm^3, unless due to disease involvement in the bone marrow
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior therapeutic intervention with any of the following:

  * Therapeutic anticancer antibodies within 4 weeks (rituximab), except within 6 months for obinutuzumab or a similar investigational type II monoclonal antibody;
  * Radio- or toxin-immunoconjugates within 10 weeks;
  * Inhibitors of BTK (ibrutinib), PI-3K (idelalisib), BH3-mimetic venetoclax, lenalidomide and other "targeted" therapy (including but not limited to investigational BTK and PI-3K inhibitors, etc.) - within 6 half-lives (i.e., 36 hours for ibrutinib)
  * All other chemotherapy, radiation therapy within 3 weeks prior to initiation of therapy
  * SYK inhibitors at any time
* Inadequate recovery from adverse events related to prior therapy to grade =< 1 (excluding grade 2 alopecia and neuropathy)
* Chronic use of corticosteroids in excess of prednisone 30 mg/day or its equivalent
* Stem cell transplant recipients must have no evidence of and not receive treatment for graft-versus-host disease
* Concomitant use or use in the prior two weeks of moderate or strong CYP3A and CYP2C9 inducers or strong CYP2C9 inhibitors, including nutraceutical preparations, e.g., grapefruit juice and St John's wort
* History prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of therapy on current study
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease
  * Adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease
  * Asymptomatic prostate cancer managed with "watch and wait" strategy
  * Myelodysplastic syndrome which is clinically well controlled and no evidence of the cytogenetic abnormalities characteristic of myelodysplasia on the bone marrow at screening
* Uncontrolled immune hemolysis or thrombocytopenia (positive direct antiglobulin test in absence of hemolysis or history of immune-mediated cytopenias are not exclusions)
* History of human immunodeficiency virus (HIV) infection or active hepatitis B or C
* Major surgery (requiring general anesthesia) within 2 weeks prior to initiation of therapy
* Inability to swallow and retain an oral medication; patients with clinically significant medical condition of malabsorption, inflammatory bowel disease, chronic conditions which manifest with diarrhea, refractory nausea, vomiting or any other condition that will interfere significantly with drug absorption are excluded; patients must also have adequate venous access
* Need for ongoing therapy with proton pump inhibitors; H2 antagonists are allowed
* Active uncontrolled infection
* Women who are pregnant or lactating
* Fertile men or women of childbearing potential unless 1) permanently sterile or 2) using a highly effective measure of contraception such as condoms in males and consistent and correct use of one of the following in females: intrauterine device, tubal sterilization, Essure micro-insert system, vasectomy in the male partner; effective contraception is required for males during treatment with study drug and to continue for 3 months after the last dose of either entospletinib or obinutuzumab, whichever is later; for women, effective contraception is required to continue for 18 months after the last dose of obinutuzumab or for 30 days after the last dose of entospletinib, whichever is later

  * Definition of childbearing potential: for this study, a female subject is considered of childbearing potential until becoming post-menopausal unless permanently sterile or with medically documented ovarian failure; women are considered to be in a postmenopausal state when >= 54 years of age with cessation of previously occurring menses for >= 12 months without an alternative cause; women of any age with amenorrhea of >= 12 months may also be considered post-menopausal if their follicle stimulating hormone (FSH) level is in the post-menopausal range and they are not using hormonal contraception or hormonal replacement therapy; permanent sterilization in females includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy in a female subject of any age; permanent sterilization in males include bilateral orchiectomy or medical documentation of alternative explanation
* Any condition for which participation in the study is judged by the Investigator to be detrimental to the patient with inter-current illness or psychiatric/social situations that would jeopardize compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Okada, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Consensus resolution: proposed criteria for evaluation of response to treatment in hairy cell leukemia. Leukemia. 1987 Apr;1(4):405. No abstract available. PMID 3669765
- [Derived] Lam V, Best S, Kittai A, Orand K, Spurgeon SE, Liu T, Danilov AV. Proapoptotic and immunomodulatory effects of SYK inhibitor entospletinib in combination with obinutuzumab in patients with chronic lymphocytic leukaemia. Br J Clin Pharmacol. 2022 Feb;88(2):836-841. doi: 10.1111/bcp.14962. Epub 2021 Jul 19. PMID 34196037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One (1) participant was initially enrolled onto the study Dose Escalation phase, but was removed from study due to subsequent discovery of transformed disease at the time of screening. This participant is not included in safety nor efficacy analysis sets.
Groups:
- Phase 1, Dose 1: Received entospletinib at Dose Level 1: 400 mg daily (200 mg twice daily) in combination with obinutuzumab during Dose Escalation phase of study.
- Phase 1, Dose 2: Received entospletinib at Dose Level 2: 800 mg daily (400 mg twice daily) in combination with obinutuzumab during Dose Escalation phase of study.
- Phase 2, MTD: Received entospletinib at Maximum Tolerated Dose (MTD) in combination with obinutuzumab during Dose Expansion phase of study.
  The MTD was determined to be 800 mg daily (400 mg twice daily).
Period: Stage 1 - Dose Escalation
Arm/Group | Phase 1, Dose 1 | Phase 1, Dose 2 | Phase 2, MTD
Started | 6 | 3 | 0
Completed | 6 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Stage 2 - Dose Expansion
Arm/Group | Phase 1, Dose 1 | Phase 1, Dose 2 | Phase 2, MTD
Started | 0 | 0 | 15
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1, Dose 1 | Phase 1, Dose 2 | Phase 2, MTD | Total
Number analyzed (Participants) | 6 | 3 | 14 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 0 | 4 | 8
  >=65 years | 2 | 3 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.03 (15.67) | 68.03 (3.82) | 67.07 (8.22) | 65.62 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 5 | 6
  Male | 5 | 3 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 6 | 2 | 10 | 18
  Unknown or Not Reported | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 1 | 12 | 19
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Entospletinib in Combination With Obinutuzumab
Description: The dose of obinutuzumab remains fixed in standard doses while the dose of entospletinib will be escalated. The starting dose of entospletinib will be 200 mg (twice-daily) and escalated to the second dose level 400 mg (twice-daily). MTD is the dose associated with a total of 6 patients treated with less than 2 dose limiting toxicities (DLT), or a total of 3 patients treated with less than 1 DLT. DLT is defined as 1) grade 3 or higher non-hematological toxicity (except grade 3 nausea, vomiting or diarrhea that was reversible within 72 hours with supportive care; grade 3 infusion-related toxicity; asymptomatic grade 3-4 laboratory abnormalities that are reversible to grade 2 or less within 72 hours; grade 3 tumor lysis syndrome or hyponatremia); 2) grade 4 neutropenia lasting >7 days or febrile neutropenia; or 3) grade 4 thrombocytopenia/anemia or grade 3 thrombocytopenia with bleeding. The dosage follows the 3+3 traditional escalation rules.
Time Frame: Up to 28 days
Measure: Number; unit: mg orally twice-daily
Groups:
- Phase 1, Dose 1-2: 2 groups of patients in phase 1 study.
  Phase 1, Dose 1 received entospletinib at Dose Level 1: 400 mg daily (200 mg twice daily) in combination with obinutuzumab during Dose Escalation phase of study. Phase 1, Dose 2 received entospletinib at Dose Level 2: 800 mg daily (400 mg twice daily) in combination with obinutuzumab during Dose Escalation phase of study.
Arm/Group | Phase 1, Dose 1-2
Number analyzed (Participants) | 9
mg orally twice-daily | 400

2. Primary Outcome: Complete Response (CR) Defined as the Percentage of Subjects Who Achieve CR
Description: Response for CLL/SLL measured using Modified International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 (IWCLL) guidelines. Response for hairy cell leukemia was measured using Consensus resolution: proposed criteria published in Leukemia 1987.
Time Frame: Up to 45 months
Population: Efficacy evaluable population: participants with CLL (Phase I/Phase II)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Research Participants: The Outcome Measure was assessed in aggregate, combining participants from both phases of the study, as per the planned protocol.
  Phase 1, Dose 1 received entospletinib at Dose Level 1: 400 mg daily (200 mg twice daily) in combination with obinutuzumab during Dose Escalation phase of study.
  Phase 1, Dose 2 received entospletinib at Dose Level 2: 800 mg daily (400 mg twice daily) in combination with obinutuzumab during Dose Escalation phase of study.
  Phase 2, MTD: Received entospletinib at Maximum Tolerated Dose (MTD) in combination with obinutuzumab during Dose Expansion phase of study. The MTD was determined to be 800 mg daily (400 mg twice daily).
Arm/Group | All Research Participants
Number analyzed (Participants) | 21
percentage of participants | 14.3 [3.0 to 36.3]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Defined as percentage of participants with complete remission, complete response with incomplete marrow recovery, partial remission and nodular partial response. Response for CLL/SLL measured using Modified International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 (IWCLL) guidelines. Response for hairy cell leukemia was measured using Consensus resolution: proposed criteria published in Leukemia 1987.
Time Frame: Up to 45 months
Population: Efficacy evaluable population: participants with CLL (Phase I/Phase II)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Research Participants
Number analyzed (Participants) | 21
Percentage of participants | 66.7 [43.0 to 85.4]

4. Secondary Outcome: Event Free Survival (EFS)
Description: Will be summarized descriptively using the Kaplan-Meier estimate. EFS will be censored if entospletinib is discontinued for other reasons (such as drug is no longer available).
Time Frame: The interval between the date of first study treatment and the date of objective signs of disease recurrence, subsequent anti leukemic therapy, or death, whichever is first reported, assessed up to 45 months.
Population: Efficacy evaluable population: participants with CLL (Phase I/Phase II)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Research Participants
Number analyzed (Participants) | 21
Months | 24.0 [16 to 28]

5. Secondary Outcome: Number of Participants Who Experienced Adverse Events
Description: Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Will be summarized for the safety population separately for phase 1 and phase 2 portions by dose level. All adverse events (AEs) will be coded by system organ class, Medical Dictionary for Regulatory Activities (MedDRA) preferred term, and severity grade using NCI CTCAE (version 4.03).
Time Frame: Up to 45 months
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1, Dose 1 (400 mg Entospletinib Daily): Patients receive entospletinib PO either QD or BID on days -7 to -1 (run-in phase) according to dose level 1 (200 mg twice daily). Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of the first cycle, and on day 1 of subsequent cycles. Treatment with obinutuzumab repeats every 28 days for up to 6 cycles and daily treatment with entospletinib continues every 28 days for up to 12 cycles in the absence of disease progression or unexpected toxicity.
  Entospletinib: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Obinutuzumab: Given IV
  Pharmacological Study: Correlative studies
- Phase 2 and MTD (800 mg Entospletinib Daily): Patients receive entospletinib PO either QD or BID on days -7 to -1 (run-in phase) according to dose level 2 (400 mg twice daily). Patients also receive obinutuzumab IV on days 1, 2, 8 and 15 of the first cycle, and on day 1 of subsequent cycles. Treatment with obinutuzumab repeats every 28 days for up to 6 cycles and daily treatment with entospletinib continues every 28 days for up to 12 cycles in the absence of disease progression or unexpected toxicity. Entospletinib is administered PO.
Arm/Group | Phase 1, Dose 1 (400 mg Entospletinib Daily) | Phase 2 and MTD (800 mg Entospletinib Daily)
Number analyzed (Participants) | 6 | 17
Participants | 6 | 17

6. Other Pre Specified Outcome: Peripheral Blood B-cell Depletion and Recovery
Description: Will be summarized using descriptive statistics.
Time Frame: Up to 45 months
Population: Data for this outcome was not collected due to PI transition.
Arm/Group | All Research Participants
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Pharmacodynamics Parameters of NFkappaB Activation and Expression of Anti-apoptotic Proteins in Chronic Lymphocytic Leukemia (CLL) Cells
Description: Pharmacokinetic parameters including peak and trough levels will be determined by noncompartmental method(s) using the pharmacokinetic profile of entospletinib and obinutuzumab.
Time Frame: Up to 45 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Biomarkers (Chromosomal Abnormalities, IGHV Mutational Status, p53 Mutational Status)
Description: Will be assessed by IgH somatic hypermutation assay version 2.0. Will associate with response (ORR) to entospletinib (ENTO) in combination with obinutuzumab in patients with relapsed/refractory CLL.
Time Frame: Up to 45 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 45 months. For the participants, the median follow-up time for adverse events was 17 months.
Description: Per protocol; "Safety data will be summarized for the safety population separately for phase 1 and phase 2 portions by dose level. All AEs will be coded by system organ class, MedDRA preferred term, and severity grade using NCI CTCAE (v 4.03)." Since Phase 2 and the subset of Phase I patients who received MTD both received 800 mg daily, these are reported together. Those who received 400 mg daily were reported separately.
Groups:
- Phase 1, Dose 1 (400 mg Entospletinib Daily): Patients receive entospletinib PO either QD or BID on days -7 to -1 (run-in phase) according to dose level 1 (200 mg twice daily). Patients also receive obinutuzumab IV on days 1, 2, 8, and 15 of the first cycle, and on day 1 of subsequent cycles. Treatment with obinutuzumab repeats every 28 days for up to 6 cycles and daily treatment with entospletinib continues every 28 days for up to 12 cycles in the absence of disease progression or unexpected toxicity.
- Phase 2 and MTD (800 mg Entospletinib Daily): Patients receive entospletinib PO either QD or BID on days -7 to -1 (run-in phase) according to dose level 2 (400 mg twice daily). Patients also receive obinutuzumab IV on days 1, 2, 8 and 15 of the first cycle, and on day 1 of subsequent cycles. Treatment with obinutuzumab repeats every 28 days for up to 6 cycles and daily treatment with entospletinib continues every 28 days for up to 12 cycles in the absence of disease progression or unexpected toxicity.
Arm/Group | Phase 1, Dose 1 (400 mg Entospletinib Daily) | Phase 2 and MTD (800 mg Entospletinib Daily)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/17
Serious Adverse Events (participants affected / at risk) | 3/6 | 5/17
Other Adverse Events (participants affected / at risk) | 6/6 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose 1 (400 mg Entospletinib Daily) (N=6) | Phase 2 and MTD (800 mg Entospletinib Daily) (N=17)
Infusion Related Reaction (General disorders) | 2 (2) | 1 (1)
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Interoperative Hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — SARS-COV2 Infection
Febrile neutropenia (Investigations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — Pneumonia
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1, Dose 1 (400 mg Entospletinib Daily) (N=6) | Phase 2 and MTD (800 mg Entospletinib Daily) (N=17)
Alanine aminotransferase increased (Investigations) | 2 (3) | 4 (11)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 5 (13)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 11 (13)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (10) | 10 (45)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 5 (13)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 3 (6)
Tooth infection (Infections and infestations) | 0 (0) | 2 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2) | 7 (17)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03010358/Prot_SAP_000.pdf